CLINICAL TRIAL: NCT04440046
Title: Real Versus Sham Manual Therapy in Addition to Therapeutic Exercise in the Treatment of Rotator Cuff Related Shoulder Pain: a Randomized Controlled Trial
Brief Title: Real Versus Sham Manual Therapy for RCRSP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alcala (Other)
Responsible Party: Principal Investigator, Prof. Dr. Daniel Pecos Martín, Principal Investigator, University of Alcala
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2/111/729
Record Dates: First submitted 2020-06-15; First posted 2020-06-19 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Shoulder Pain
MeSH Terms: conditions — Shoulder Pain | interventions — Exercise Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Real manual therapy (Experimental): Real manual therapy directed to the thoracic spine and glenohumeral joint added to a therapeutic exercise program
  Interventions: Other: Manual therapy thoracic spine; Other: Manual therapy glenohumeral joint; Other: Therapeutic exercise
- Sham thoracic manual therapy (Sham Comparator): Sham manual therapy directed to the thoracic spine with real manual therapy directed to the glenohumeral joint added to the same therapeutic exercise program performed in the real manual therapy group
  Interventions: Other: Manual therapy glenohumeral joint; Other: Sham thoracic manual therapy; Other: Therapeutic exercise
- Sham manual therapy (Sham Comparator): Sham manual therapy directed to the thoracic spine and glenohumeral joint added to the same therapeutic exercise program performed in the real manual therapy group
  Interventions: Other: Sham thoracic manual therapy; Other: Sham glenohumeral manual therapy; Other: Therapeutic exercise

INTERVENTIONS:
Other: Manual therapy thoracic spine — Manual therapy mobilization directed to the costovertebral joint.
  Arms: Real manual therapy
Other: Manual therapy glenohumeral joint — Manual therapy mobilization directed to the glenohumeral joint.
  Arms: Real manual therapy; Sham thoracic manual therapy
Other: Sham thoracic manual therapy — Sham manual therapy directed to the costovertebral joint.
  Arms: Sham manual therapy; Sham thoracic manual therapy
Other: Sham glenohumeral manual therapy — Sham manual therapy directed to the glenohumeral joint.
  Arms: Sham manual therapy
Other: Therapeutic exercise — Therapeutic exercise program consisting on isometric exercise with progressive load.

SUMMARY:
A convenience sample of subjects with RCRSP recruited through announcements at the Benemerita Universidad Autonoma de Puebla will be treated with an exercise program with sham or real manual therapy for 5 weeks.

The hypothesis of the present study is that the addition of manual therapy to a therapeutic exercise program produces better benefits in comparison to the same exercise program with sham manual therapy procedures in the management of patients with RCRSP.

DETAILED DESCRIPTION:
The objective of this study is to demonstrate that the combination of manual therapy and therapeutic exercise achieves better results in the management of the patient with shoulder pain.

For this, manual therapy techniques in the thoracic region and in the shoulder together with a therapeutic exercise program will be applied.

The investigators will compare this intervention protocol with placebo manual therapy techniques and the same therapeutic exercise protocol.

ELIGIBILITY:
Inclusion Criteria:

* unilateral shoulder pain of non-traumatic origing lasting more than three months.
* Pain evoked with active shoulder movements.
* Pain and weakness evoked with manual muscle strength tests for abduction and/or external rotation.
* Minimal or no rest pain (less than 3 points in a numeric pain rating scale).

Exclusion Criteria:

* Other shoulder pathologies than RCRSP.
* Systemic diseases.
* Neural symptoms.
* Neck pain.
* Radiculopathy.
* To have been treated for shoulder pain in the last three months.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2020-12-15 (Actual); Primary Completion 2021-04-18 (Actual); Study Completion 2021-04-18 (Actual)

PRIMARY OUTCOMES:
Shoulder Pain and Disability Index (SPADI) | Change from Baseline at 17- week
  The SPADI points from 0 (no disability) to 130 (maximum degree of disability)

SECONDARY OUTCOMES:
Pain intensity measured with a visual analogue scale | Change from Baseline at 17-week
  10-cm scale where 0 is no pain and 10 is the worst pain imaginable
Pain-free range of movement of the shoulder | Change from Baseline at 17-week
  Flexion, extension, abduction, internal rotation and external rotation measured with a two-arm goniometer

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Pecos-Martin, PhD, Study Director — University of Alcala
Locations (1):
- Ruben Fernandez-Matias, Alcalá de Henares, Spain

IPD SHARING:
Plan to Share IPD: No